CLINICAL TRIAL: NCT04228952
Title: STUDY 2: CLINICAL PROTOCOL Metabolism of NNK Among Japanese Americans
Brief Title: Metabolism of NNK in Japanese Americans
Status: Completed | Type: Observational
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: University of Hawaii (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2019NTUC208; P01CA138338 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Smoking
Keywords: CYP2A6, Nicotine Metabolite Ratio, NNAL, NNK α-hydroxylation
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 24 hour urine and blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smokers with very low or no CYP2A6 activity: Japanese American smokers (daily > 5 cigarettes) with little or no CYP2A6 activity (CYP2A6 activity defined as a ratio of trans-3-hydroxycotinine:cotinine ratio of <0.6).
  Interventions: Combination Product: Modified Natural American Spirit-Tan or Green cigarettes injected with labeled NNK
- Smokers with high CYP2A6 activity: Japanese American smokers (daily > 5 cigarettes) with high CYP2A6 activity (CYP2A6 activity defined as a ratio of trans-3-hydroxycotinine:cotinine ratio of > 3.0)
  Interventions: Combination Product: Modified Natural American Spirit-Tan or Green cigarettes injected with labeled NNK

INTERVENTIONS:
Combination Product: Modified Natural American Spirit-Tan or Green cigarettes injected with labeled NNK — American Spirit cigarettes will be modified by adding 0.300 μg [pyridine-D4]NNK to each cigarette so that the amount of total (deuterated plus unlabeled) NNK in these cigarettes is below 0.700 μg/g tobacco.

SUMMARY:
The risk of lung cancer varies by individual and by ethnic/racial group. In this study the investigators will explore how individual differences in the metabolism of a tobacco-specific lung carcinogen may contribute to the variable risk of lung cancer between ethnic/racial groups.

In this 10 day clinical trial, Japanese Americans will smoke a cigarette containing deuterium-labeled 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK), a tobacco-specific lung carcinogen. The study cigarette will be smoked for 7 days.

This will allow for NNK metabolic profiling and determining the effect of CYP2A6 genotype on the level of NNK α-hydroxylation in Japanese Americans smokers using [pyridine- D4]-NNK containing cigarettes.

DETAILED DESCRIPTION:
Eligible subjects will provide a baseline 24 hour urine sample. Study cigarettes spiked with labeled NNK will be provided to the subjects to smoke over a 7 day period. During this time, 24 hour urine samples will be collected over days 5, 6 and 7 on study cigarettes. Blood will be drawn on days 6 and 7 on study cigarettes. Samples will be analyzed for NNK metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese American - one, but preferably 2 biological parents of Japanese descent
2. 21 years or older
3. Daily smoker
4. Eligible urinary ratios of total 3-hydroxycotinine to cotinine (3HC/COT):

   * "Little or no-CYP2A6 activity" defined as a 3-hydroxycotinine:cotinine ratio of <0.6 or
   * "Relatively high" CYP2A6 activity defined as a 3-hydroxycotinine:cotinine ratio of >3.0.
5. Stable and good physical and mental health
6. Provided written informed consent to participate in the study

Exclusion Criteria:

1. Unwilling to avoid other nicotine containing products during the study and no use of any nicotine-containing products except cigarettes for 1 week prior to their study visits
2. Currently taking any medications that affect relevant metabolic enzymes
3. Experiencing medical conditions that might affect biomarkers of exposure and effect
4. Pregnant or nursing or planning on becoming pregnant during the study
5. Unable to read and understand English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Japanese American Smokers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2025-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Hatsukami, Ph.D, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available in two formats: Summary of the data (graphs and tables) and as raw individual-level data for analysis. Requests for data must be in writing, identify the affiliation and describe how the data will be used. Users agree not to transfer the data to other users and that the data are only to be used for research purposes. The PI will require requestors of data to sign a data and biospecimen sharing agreement that will ensure (1) Use of only for research purposes and not to identify any individual or personal information, (2) Data will be secure, (3) Destruction or return of data after data analysis and (4) Proper citation in publications or other written materials. A record of transfer of data and a copy of the dataset that was distributed will be kept by University of Minnesota.
Time Frame: Data will be available after papers are accepted for publication
Access Criteria: Data generated by this grant will be made to outside investigators, according to the Guidance at http://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smokers With Very Low or no CYP2A6 Activity | Smokers With High CYP2A6 Activity
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smokers With Very Low or no CYP2A6 Activity | Smokers With High CYP2A6 Activity | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Ratio of D4-hydroxy Acid to D4- NNAL (an Estimate if NNK Alpha Hydroxylation)
Description: Difference in means of the ratio of D4-hydroxy acid to D4- NNAL (an estimate if NNK alpha hydroxylation) for the two groups (null versus average CYP2A6 activity)
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Smokers With Very Low or no CYP2A6 Activity | Smokers With High CYP2A6 Activity
Number analyzed (Participants) | 8 | 8
Ratio | 0.133 (0.096) | 0.175 (0.066)

ADVERSE EVENTS:
Time Frame: 1 days
Arm/Group | Smokers With Very Low or no CYP2A6 Activity | Smokers With High CYP2A6 Activity
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT04228952/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT04228952/ICF_001.pdf